CLINICAL TRIAL: NCT06429943
Title: Cerebrolysin in Patients Diagnosed With SAH - an Observational Cohort Study (PILOT)
Brief Title: Cerebrolysin in SAH (Subarachnoidal Haemorrhage) - Observational Study
Status: Completed | Type: Observational
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Sponsor
Other Study IDs: SAH/2020/2023
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2023-12

CONDITIONS: SAH (Subarachnoid Hemorrhage)
Keywords: SAH; Cerebrolysin; neuromonitoring
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- A: Cerebrolysin administration
- B: without Cerebrolysin administration

SUMMARY:
Subarachnoid haemorrhage often affects people in middle age and is associated with high mortality or neurological damage. In recent years, advances in surgical techniques have im-proved the mortality rate. However, there is still need for the research for the optimal possible final effect of treatment. In our study, we've decided to examine the effect of a multimodal approach including Cerebrolysin in the supportive treatment of patients. We've examined the supply of neuroprotective drugs and neuromonitoring.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years old, diagnosis of SAH, treatment in ICU conditions

Exclusion Criteria:

* age <18 years, medical history of allergy to Cerebrolysin, acute renal failure, pregnancy, multi organ trauma, death within 48 hours after admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is the population of patients diagnosed with SAH, treated in University Hospital no.1 in Szczecin, Poland. Mainly the patients come from the population of westerpomeranian county, but as SAH is an acute disease also patients from the whole region of Poland, treated in the Hospital were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
GOS Glasgow Outcome Scale | 1 month
  Glasgow Outcome Scale - 5 points scale, characterizing the patients' deficits

SECONDARY OUTCOMES:
LOS Length of Stay | hospitalisation time
  length of stay in days, that patient spent in hospital/ intensive care unit
mortality | 1 month
  mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Pomeranian Medical University, University Hospital no.1, Szczecin, Poland